CLINICAL TRIAL: NCT02414958
Title: A Phase III, Randomised, Double Blind, Placebo-controlled, Parallel Group, Efficacy, Safety and Tolerability Trial of Once Daily, Oral Doses of Empagliflozin as Adjunctive to inSulin thErapy Over 52 Weeks in Patients With Type 1 Diabetes Mellitus (EASE-2)
Brief Title: Empagliflozin as Adjunctive to InSulin thErapy Over 52 Weeks in Patients With Type 1 Diabetes Mellitus (EASE-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.69; 2014-001922-14 (EudraCT Number)
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — empagliflozin

ARMS (3):
- Empagliflozin low dose (Experimental): Empagliflozin tablets once daily
  Interventions: Drug: Empagliflozin
- Empagliflozin high dose (Experimental): Empagliflozin tablets once daily
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): Placebo tablets matching empagliflozin once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin
  Arms: Empagliflozin low dose
Drug: Empagliflozin
  Arms: Empagliflozin high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Comparison of 2 doses of empagliflozin vs placebo in patients already using either an insulin regimen of multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII). Randomisation to 3 treatments arms (equal assignment) following a screening period, an optimisation period and a run-in period. 52 week double-blind treatment period, and 3 week follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Male or female patient receiving insulin for the treatment of documented diagnosis of Type 1 Diabetes Mellitus (T1DM) for at least 1 year at the time of Visit 1
* Fasting C-peptide value of < 0.7 ng/mL (0.23 nmol/L) at Visit 2 measured by the central laboratory
* Use of, and be willing, based on the Investigator's judgement, to continue throughout the duration of the trial, either:

  * Multiple Daily Injections (MDI) of insulin consisting of at least one basal insulin injection and at least three daily bolus injections OR
  * Continuous Subcutaneous Insulin Infusion (CSII) of any insulin type, with at least 5 months experience of using CSII prior to Visit 1
* HbA1c >/= 7.5% and </= 10.0% at Visit 5 measured by the central laboratory
* Age >/= 18 years at Visit 1

Additional inclusion criteria may apply

Exclusion criteria:

* History of Type 2 Diabetes Mellitus (T2DM), maturity onset diabetes of the young (MODY), pancreatic surgery or chronic pancreatitis
* Pancreas, pancreatic islet cells or renal transplant recipient
* T1DM treatment with any other antihyperglycaemic drug (e.g. metformin, alpha-glucosidase inhibitors, Glucagon-like-peptide 1 (GLP-1) analogues, Sodium-Glucose Co-Transporter (SGLT-2) inhibitors, pramlintide, inhaled insulin, pre-mixed insulins etc.) except subcutaneous basal and bolus insulin within 3 months prior to Visit 1
* Occurrence of severe hypoglycaemia involving coma/unconsciousness and/or seizure that required hospitalisation or hypoglycaemia-related treatment by an emergency physician or paramedic within 3 months prior to Visit 1 and until randomisation
* Occurence of Diabetic Ketoacidosis (DKA) within 3 months prior to Visit 1 and until randomisation

Additional exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (131):
- United States (34):
  - AMCR Institute, Inc., Escondido, California
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - National Research Institute, Los Angeles, California
  - Mills-Peninsula Health Services, San Mateo, California
  - Metabolic Institute of America, Tarzana, California
  - University Clinical Investigators, Inc., Tustin, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Baptist Diabetes Associates, PA, Miami, Florida
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Northwest Endo Diabetes Research, LLC, Arlington Heights, Illinois
  - Midwest Endocrinology, Crystal Lake, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Diabetes anddocrine Associates, PC, Omaha, Nebraska
  - Desert Endocrinology Clinical Research Center, Henderson, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Albany Medical Center / Albany Medical College, Albany, New York
  - University Physicians Group Research Division, Staten Island, New York
  - Diabetes and Endocrinology Consultants, PC, Morehead City, North Carolina
  - The Carl and Edyth Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Diabetes and Obesity Clinical Trials Center, Nashville, Tennessee
  - North Texas Endocrine Center, Dallas, Texas
  - Office of Dr. Michelle Zaniewski-Singh, Houston, Texas
  - Texas Diabetes and Endocrinology, Round Rock, Texas
  - Bateman Horne Center, Salt Lake City, Utah
  - Advanced Research Institute, South Ogden, Utah
  - Larry D Stonesifer, MD Inc., PS, Federal Way, Washington
  - Rainier Clinical Research Center, Inc, Renton, Washington
  - The Polyclinic, Seattle, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Australia (3):
  - Coffs Endocrine & Diabetes Services, Coffs Harbour, New South Wales
  - AIM Centre, Merewether, New South Wales
  - Royal Brisbane & Women's Hospital-Endocrinology, Herston, Queensland
- Austria (4):
  - VIVIT Instit.am LKH Feldkirch,Abt.f.Innere Med.u.Kardiologie, Feldkirch
  - LKH Steyr, Kardiologie, Steyr
  - KH Rudolfstiftung, 1. Med. Abt., Wien, Vienna
  - Hospital Hietzing, Vienna
- Belgium (11):
  - Arlon - HOSP Sud Luxembourg - Vivalia, Arlon
  - Bonheiden - HOSP Imelda, Bonheiden
  - ULB Hopital Erasme, Brussels
  - Brussels - UNIV UZ Brussel, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UNIV UZ Gent, Ghent
  - La Louvière - UNIV CHU Tivoli, La Louvière
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Liège - HOSP CHR de la Citadelle, Liège
  - Merksem - HOSP ZNA Jan Palfijn, Merksem
- Canada (10):
  - LMC Endocrinology Centres (Calgary) Ltd., Calgary, Alberta
  - The Bailey Clinic, Red Deer, Alberta
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Health Sciences Centre Winnipeg, Winnipeg, Manitoba
  - CHUM - Pavillon R, Montreal, Migration Data
  - Capital District Health Auth., Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - LMC Thornhill/Vaughan, Thornhill, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- Czechia (3):
  - General Univ.hosp.in Prague (VFN), Diabetes ambulance, Prague
  - Diabetology and Internal Practice Dr. Vladimir Lelek, Slaný
  - Masaryk Hospital, Internal Department, Ústí nad Labem
- Denmark (5):
  - Aalborg Sygehus Syd, Aalborg
  - Aarhus Universitets Hospital, Aarhus C
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Nordsjællands Hospital - Hillerød, Hillerød
  - Køge Sygehus, Køge
- Finland (3):
  - IteLasaretti, Kuopio
  - Terveystalo Oulu, Diapolis, Oulu
  - TYKS, Turku
- France (6):
  - HOP Côte de Nacre, Caen
  - HOP Saint-Louis, La Rochelle
  - HOP de Narbonne, diabéto endo, Narbonne, Narbonne
  - HOP Robert Debré, Reims
  - HOP de Brabois, Vandœuvre-lès-Nancy
  - HOP les Portes du Sud, Diabéto, Vénissieux, Vénissieux
- Germany (9):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Gemeinschaftspraxis, Asslar, Aßlar
  - ikfe - Institut für klinische Forschung und Entwicklung Berlin GmbH, Berlin
  - InnoDiab Forschung GmbH, Essen
  - Praxis Dr. Kosch, Pirna, Pirna
  - Allgemeinmedizinische und Diabetologische Schwerpunktpraxis, Rehlingen-Siersburg
  - Praxis Dr. Hirschhäuser, Saarbrücken
  - Praxis Dr. Segner, St. Ingbert, Saint Ingbert/Oberwürzbach
  - Ambulanzzentrum Schweinfurt, Schweinfurt
- Netherlands (7):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Rijnstate Hospital, Arnhem
  - Martini Ziekenhuis, Groningen
  - Bethesda Ziekenhuis Hoogeveen, Hoogeveen
  - Sint Franciscus Gasthuis, Rotterdam
  - Albert Schweitzer Ziekenhuis, Zwijndrecht, Zwijndrecht
- Norway (4):
  - Helse Møre og Romsdal HF, Ålesund sjukehus, Ålesund
  - Sykehuset Innlandet HF, Avd. Hamar, Hamar
  - Akershus Universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF, Aker Sykehus, Oslo
- Poland (8):
  - Med Univ Bialystok Clin Dep Endocrinol, Diabetol & Int Dis, Bialystok
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny, Bialystok
  - Dobry Lekarz,Spec.Med.Clinics,Private Prac,Krakow, Krakow
  - NZOZ Specialized Ambulance "MEDICA", Lublin
  - Marcinkowski Poznan Univ of Med Sci, Clin Dept Diab, Poznan, Poznan
  - NZOZ Centrum Medyczne AESKULAP,Private Prac, Radom, Radom
  - Centrum Medyczne Medyk, Rzeszów
  - NBR Polska, Warsaw
- Spain (7):
  - C.A.P. Sardenya, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de la Inmaculada Concepción, Granada
  - Hospital Virgen de la Victoria, Málaga
  - Hospital General de Segovia, Segovia
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Virgen Macarena, Seville
- Sweden (3):
  - Ladulaas Kliniska Studier, Borås
  - Centralsjukhuset, Karlstad, Karlstad
  - Läkarhuset, Vällingby, Vällingby
- Taiwan (5):
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- United Kingdom (9):
  - Milton Keynes Hospital, Buckinghamshire
  - Addenbrooke's Hospital, Cambridge
  - Wellcome Trust Clinical Research Facility, Edinburgh
  - Leicester General Hospital, Leicester
  - Royal London Hospital, London
  - Queen's Medical Centre, Nottingham
  - George Eliot Hospital, Nuneaton
  - East Surrey Hospital, Surrey
  - Queen Elizabeth II Hospital, Welwyn Garden City

REFERENCES:
- [Derived] Song C, Dhaliwal S, Bapat P, Scarr D, Bakhsh A, Budhram D, Verhoeff NJ, Weisman A, Fralick M, Ivers NM, Cherney DZI, Tomlinson G, Lovblom LE, Mumford D, Perkins BA. Point-of-Care Capillary Blood Ketone Measurements and the Prediction of Future Ketoacidosis Risk in Type 1 Diabetes. Diabetes Care. 2023 Nov 1;46(11):1973-1977. doi: 10.2337/dc23-0840. PMID 37616393
- [Derived] Rosenstock J, Marquard J, Laffel LM, Neubacher D, Kaspers S, Cherney DZ, Zinman B, Skyler JS, George J, Soleymanlou N, Perkins BA. Empagliflozin as Adjunctive to Insulin Therapy in Type 1 Diabetes: The EASE Trials. Diabetes Care. 2018 Dec;41(12):2560-2569. doi: 10.2337/dc18-1749. Epub 2018 Oct 4. PMID 30287422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, double-blind, placebo-controlled, parallel group, 52-week trial comparing 2 oral once daily doses (10 mg and 25 mg) of empagliflozin with placebo in patients with type 1 diabetes mellitus (T1DM), each as adjunctive to optimised insulin therapy.
Pre-assignment Details: 6-week T1DM therapy (insulin) optimisation period followed by a 2-week placebo run-in period before randomisation. Patients who successfully completed both of the periods were randomised into the 52-week double-blind treatment period. All treatments were administered in addition to optimised insulin therapy.
Groups:
- Placebo Matching Empagliflozin: Patients administered placebo matching empagliflozin film-coated tablet orally once daily as adjunctive to optimised insulin therapy for 52 weeks
- Empagliflozin 10 mg: Patients administered empagliflozin 10 mg film-coated tablet orally once daily as adjunctive to optimised insulin therapy for 52 weeks.
- Empagliflozin 25 mg: Patients administered empagliflozin 25 mg film-coated tablet orally once daily as adjunctive to optimised insulin therapy for 52 weeks.
Period: Overall Study
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 243 | 243 | 244
Completed | 211 | 223 | 230
Not Completed | 32 | 20 | 14
Not completed — Adverse Event | 6 | 6 | 3
Not completed — Protocol Violation | 10 | 3 | 1
Not completed — Lost to Follow-up | 7 | 4 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 5
Not completed — Other than specified | 4 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Randomised set (RS): All patients from the screened set (SCR) who were randomised to trial medication regardless of whether any trial medication was taken.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 243 | 243 | 244 | 730
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: RS
  Years | 44.2 (13.6) | 45.7 (12.5) | 45.3 (14.0) | 45.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: RS
  Participants
    Female | 133 | 125 | 131 | 389
    Male | 110 | 118 | 113 | 341
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: RS
  Participants
    Hispanic or Latino | 7 | 4 | 6 | 17
    Not Hispanic or Latino | 236 | 239 | 238 | 713
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: RS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 7 | 6 | 10 | 23
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
    Black or African American | 7 | 6 | 4 | 17
    White | 227 | 230 | 230 | 687
    More than one race | 2 | 0 | 0 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Haemoglobin (HbA1c) at Week 26
Description: Change from baseline in glycated haemoglobin (HbA1c) for full analysis set (FAS) (observed cases [OC]) is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomised trial medication. Least squares mean is adjusted mean change from baseline. Restricted maximum likelihood estimation based on mixed-effect model for repeated measures (MMRM) analysis was used to obtain adjusted means for the treatment effects.
Time Frame: Baseline to week 26
Population: Full analysis set (FAS) (observed cases [OC]): Patients in the Treated Set (TS) who had a baseline and at least 1 on-treatment HbA1c measurement; the FAS was the basis for the primary efficacy analysis
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
Percentage (%) | 0.09 (0.04) | -0.44 (0.04) | -0.44 (0.04)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; Model Mixed effect Model Repeated Measures (MMRM) included the fixed categorical effects of treatment, pre-existing insulin therapy, visit , and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline HbA1c, baseline estimated glomerular filtration rate (eGFR), and baseline HbA1c-by- visit interaction. Patient was included as random effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, Mixed effect Model Repeated Measures; Mean Difference (Final Values) = -0.54, 97.5% CI 2-sided [-0.66 to -0.41], Standard Error of Mean 0.06 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; Model MMRM included the fixed categorical effects of treatment, pre-existing insulin therapy, visit, and treatment-by- visit interaction, as well as the continuous, fixed covariates of baseline HbA1c, baseline eGFR, and baseline HbA1c-by- visit interaction. Patient was included as random effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = -0.53, 97.5% CI 2-sided [-0.66 to -0.41], Standard Error of Mean 0.06 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

2. Primary Outcome: Change From Baseline in Glycated Haemoglobin (HbA1c) at Week 26 for Modified Intention-to-treat Population Set (mITT) (Observed Case (OC) - All Data (AD) (OC-AD) )
Description: Change from baseline in glycated haemoglobin (HbA1c) for modified intention-to-treat population set (mITT) (observed case - all data [OC-AD]) is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomised trial medication. Least squares mean is adjusted mean change from baseline. Restricted maximum likelihood estimation based on mixed-effect model for repeated measures (MMRM) analysis was used to obtain adjusted means for the treatment effects.
Time Frame: Baseline to week 26
Population: Modified intention-to-treat set (mITT) (observed case - all data [OC-AD]): Patients in the TS who had a baseline and at least 1 post-baseline HbA1c measurement.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
Percentage (%) | 0.09 (0.04) | -0.43 (0.04) | -0.42 (0.04)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; Model MMRM includes baseline HbA1c, baseline eGFR as linear covariates and baseline pre-existing insulin therapy, treatment, visit, visit by treatment interaction, baseline HbA1c by visit interaction as fixed effects. Patient is included as random effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = -0.53, 97.5% CI 2-sided [-0.65 to -0.40], Standard Error of Mean 0.06 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = -0.51, 97.5% CI 2-sided [-0.64 to -0.39] — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

3. Secondary Outcome: Rate Per Patient-year of Investigator-reported Symptomatic Hypoglycaemia Adverse Events (AEs) With Confirmed Plasma Glucose (PG)
Description: This is a key secondary endpoint. Rate per patient-year of investigator-reported symptomatic hypoglycaemia adverse events (AEs) with confirmed plasma glucose (PG) <54 milligram per deciliter (mg/dL) (<3.0 millimoles per litre (mmol/L)) and/or severe hypoglycaemia AEs (i.e. all investigator-reported AEs that had confirmed PG <54 mg/dL [<3.0 mmol/L] with symptoms reported and all severe hypoglycaemia events that were confirmed by adjudication) is presented for (i) From week 5 to 26 and (ii) From week 1 to 26. Least squares mean is actually an adjusted event rate.
Time Frame: Week 5 to Week 26, Week 1 to Week 26
Population: FAS (OC)
Measure: Least Squares Mean (95% Confidence Interval); unit: Event per patient year
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
Event per patient year
  Week 5 to 26: number analyzed (Participants) | 238 | 243 | 239
  Week 5 to 26 | 8.92 [7.15 to 11.14] | 6.64 [5.32 to 8.28] | 6.48 [5.18 to 8.12]
  Week 1 to 26: number analyzed (Participants) | 239 | 243 | 241
  Week 1 to 26 | 9.13 [7.36 to 11.34] | 7.07 [5.70 to 8.76] | 7.15 [5.75 to 8.88]
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; For week 5 to 26, negative binomial model includes baseline rate of hypoglycaemia, baseline HbA1c, and baseline eGFR as linear covariates and baseline pre-existing insulin therapy and treatment as fixed effects. Log (time at risk [days]) was used as offset; Test type: Superiority; p = 0.0623, Negative binomial model; Adjusted Rate Ratio (%) = 0.744, 97.75% CI 2-sided [0.518 to 1.069] — Empagliflozin 10 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0480, Negative binomial model; Adjusted Rate Ratio (%) = 0.726, 97.75% CI 2-sided [0.502 to 1.501] — Empagliflozin 25 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; For week 1 to 26, negative binomial model includes baseline rate of hypoglycaemia, baseline HbA1c, and baseline eGFR as linear covariates and baseline pre-existing insulin therapy and treatment as fixed effects. Log (time at risk [days]) was used as offset; Test type: Superiority; p = 0.0972, Negative binomial model — This is a nominal p-value; Adjusted Rate Ratio (%) = 0.774, 95% CI 2-sided [0.572 to 1.048] — Empagliflozin 10 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate
Statistical Analysis 4: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.1180, MMRM — Negative binomial model; Adjusted Rate Ratio (%) = 0.782, 97.75% CI 2-sided [0.575 to 1.064] — Empagliflozin 25 milligram (mg) adjusted rate/Placebo matching Empagliflozin adjusted rate

4. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Change from baseline in body weight is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomised trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
Kilogram (kg) | -0.10 (0.21) | -2.79 (0.20) | -3.37 (0.20)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; Model MMRM includes baseline weight, baseline eGFR, baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, visit by treatment interaction, baseline weight by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = -2.69, 99.75% CI 2-sided [-3.57 to -1.80], Standard Error of Mean 0.29 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = -3.27, 99.75% CI 2-sided [-4.15 to -2.39] — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

5. Secondary Outcome: Change From Baseline in Percentage of Time Spent in Target Glucose Range From Weeks 23 to 26
Description: Change from baseline in the percentage of time spent in target glucose range of >70 to ≤180 mg/dL (>3.9 to ≤10.0 mmol/L) as determined by continuous glucose monitoring (CGM) is presented in week 23 to 26. Least squares mean is actually an adjusted event rate.
Time Frame: Week 23 to 26
Population: FAS observed cases excluding data after use of paracetamol (OC-P)
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
Percentage of time | -1.13 (0.72) | 10.73 (0.71) | 11.74 (0.70)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; The analysis of covariance (ANCOVA) model includes baseline time in the target range, baseline HbA1c, and baseline eGFR as linear covariates and baseline pre-existing insulin therapy and treatment as fixed effects; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 11.86, 99.75% CI 2-sided [8.78 to 14.93] — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 12.87, 99.75% CI 2-sided [9.81 to 15.93], Standard Error of Mean 1.01 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

6. Secondary Outcome: Change From Baseline in Interstitial Glucose Variability Based on the Interquartile Range (IQR) as Determined by CGM in Weeks 23 to 26
Description: Change from baseline in interstitial glucose variability based on the IQR as determined by CGM is presented for week 23 to 26. Least squares mean is actually an adjusted event rate.
Time Frame: Week 23 to 26
Population: FAS observed cases excluding data after use of paracetamol (OC-P)
Measure: Least Squares Mean (Standard Error); unit: milligrams (mg)/ deciliter (dL)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
milligrams (mg)/ deciliter (dL) | 1.62 (1.21) | -15.30 (1.18) | -17.41 (1.16)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; The analysis of covariance (ANCOVA) model includes model includes baseline IQR of glucose, baseline HbA1c, and baseline eGFR as linear covariates and baseline pre-existing insulin therapy and treatment as fixed effects; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -16.92, 99.75% CI 2-sided [-22.04 to -11.81], Standard Error of Mean 1.68 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -19.04, 99.75% CI 2-sided [-24.13 to -13.95], Standard Error of Mean 1.68 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

7. Secondary Outcome: Change From Baseline in Total Daily Insulin Dose (TDID) at Week 26
Description: Change from baseline in TDID is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomised trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: Unit/kilogram (U/kg)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
Unit/kilogram (U/kg) | -0.010 (0.007) | -0.102 (0.007) | -0.100 (0.007)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; Model MMRM includes baseline total daily insulin dose, baseline estimated eGFR, baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, visit by treatment interaction, baseline total daily insulin dose by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = -0.092, 99.75% CI 2-sided [-0.121 to -0.063], Standard Error of Mean 0.009 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, MMRM; Mean Difference (Final Values) = -0.090, 99.75% CI 2-sided [-0.119 to -0.062], Standard Error of Mean 0.009 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

8. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 26
Description: Change from baseline in SBP and DBP is presented. With regards to efficacy and safety endpoints, the term 'baseline' referred to the last observed measurement prior to administration of any randomised trial medication. Least squares mean is adjusted mean change from baseline.
Time Frame: Baseline to week 26
Population: FAS observed cases excluding data after change in use of anti-hypertensives (OC-H)
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 243 | 243 | 244
Millimeters of mercury (mmHg)
  SBP: number analyzed (Participants) | 238 | 243 | 238
  SBP | -0.8 (0.7) | -2.9 (0.7) | -4.5 (0.7)
  DBP: number analyzed (Participants) | 239 | 243 | 241
  DBP | -0.3 (0.5) | -1.6 (0.5) | -2.6 (0.5)
Statistical Analysis 1: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; For SBP, the model MMRM includes baseline SBP seated, baseline estimated eGFR, baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, treatment by visit interaction, baseline SBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p = 0.0397, MMRM; Mean Difference (Final Values) = -2.1, 99.75% CI 2-sided [-5.2 to 1.0], Standard Error of Mean 1.0 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 2: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; For SBP, the model includes baseline SBP seated, baseline estimated eGFR, baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, treatment by visit interaction, baseline SBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p = 0.0003, MMRM; Mean Difference (Final Values) = -3.7, 99.75% CI 2-sided [-6.8 to -0.6], Standard Error of Mean 1.0 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 3: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 10 mg; For DBP, the model MMRM includes baseline DBP seated, baseline eGFR baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, treatment by visit interaction, baseline DBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p = 0.0457, MMRM — Nominal p-value; Mean Difference (Final Values) = -1.3, 99.75% CI 2-sided [-2.7 to 0.0], Standard Error of Mean 0.7 — Mean Difference= Empagliflozin 10 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean
Statistical Analysis 4: Comparison: Placebo Matching Empagliflozin vs Empagliflozin 25 mg; For DBP, the model MMRM includes baseline DBP seated, baseline estimated eGFR, baseline HbA1c as linear covariate and baseline pre-existing insulin therapy, treatment, visit, treatment by visit interaction, baseline DBP seated by visit interaction as fixed effect. An unstructured covariance structure was used to model the within-patient measurements; Test type: Superiority; p = 0.0006, MMRM; Mean Difference (Final Values) = -2.3, 99.75% CI 2-sided [-4.3 to -0.3], Standard Error of Mean 0.7 — Mean Difference= Empagliflozin 25 milligram (mg) adjusted mean - Placebo matching Empagliflozin adjusted mean

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication until 7 days after last in-take of trial medication, up to 422 days
Description: Treated set (TS): all patients who were treated with at least one dose of randomised trial medication; the TS was the basis for safety analyses. The total number of participants at risk is based on treated set.
Groups:
- Placebo Matching Empagliflozin: Patients administered placebo matching Empagliflozin film-coated tablet orally once daily in addition as adjunctive to optimised insulin therapy for 52 weeks.
- Empagliflozin 10 mg: Patients administered Empagliflozin 10 mg film-coated tablet orally once daily in addition as adjunctive to optimised insulin therapy for 52 weeks.
- Empagliflozin 25 mg: Patients administered Empagliflozin 25 mg film-coated tablet orally once daily in addition as adjunctive to optimised insulin therapy for 52 weeks.
Arm/Group | Placebo Matching Empagliflozin | Empagliflozin 10 mg | Empagliflozin 25 mg
All-Cause Mortality (participants affected / at risk) | 0/243 | 0/243 | 0/244
Serious Adverse Events (participants affected / at risk) | 28/243 | 43/243 | 26/244
Other Adverse Events (participants affected / at risk) | 197/243 | 197/243 | 195/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching Empagliflozin (N=243) | Empagliflozin 10 mg (N=243) | Empagliflozin 25 mg (N=244)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 2
Glaucoma (Eye disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 1
Normal tension glaucoma (Eye disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Pleurisy viral (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bacterial test positive (Investigations) | 0 | 1 | 0
Blood ketone body increased (Investigations) | 0 | 1 | 0
Clostridium test positive (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 12 | 8
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 9 | 3
Ketoacidosis (Metabolism and nutrition disorders) | 2 | 4 | 2
Ketosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0 | 0
Lacunar stroke (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1 | 0
Radicular syndrome (Nervous system disorders) | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching Empagliflozin (N=243) | Empagliflozin 10 mg (N=243) | Empagliflozin 25 mg (N=244)
Diarrhoea (Gastrointestinal disorders) | 9 | 13 | 8
Nausea (Gastrointestinal disorders) | 14 | 12 | 14
Vomiting (Gastrointestinal disorders) | 12 | 19 | 12
Influenza (Infections and infestations) | 11 | 20 | 12
Nasopharyngitis (Infections and infestations) | 41 | 52 | 43
Sinusitis (Infections and infestations) | 13 | 14 | 9
Upper respiratory tract infection (Infections and infestations) | 25 | 15 | 27
Urinary tract infection (Infections and infestations) | 29 | 37 | 20
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 9 | 14
Blood ketone body increased (Investigations) | 10 | 18 | 20
Hypoglycaemia (Metabolism and nutrition disorders) | 152 | 154 | 147

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT02414958/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT02414958/SAP_001.pdf